CLINICAL TRIAL: NCT06173141
Title: Effect of Intradialytic Continuous Versus Interval Aerobic Exercises on Functional Capacity Quality of Life and in Patients With Chronic Renal Failure.
Brief Title: Effect of Intradialytic Continuous Versus Interval Aerobic Exercises on Functional Capacity in Patients With Chronic Renal Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Mousa Galeb, Lecturer at the Department of Physical Therapy for Cardiovascular /Respiratory Disorders and Geriatrics Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chronic renal failure
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Diseases
Keywords: Intradialytic cycling exercise, function capacity, hemodialysis, quality of life.
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Sixty-seven patients undergoing haemodialysis randomly be allocated into three groups, (A, B & C). Group A (low- to moderate-continuous intensity cycling exercises, group B (moderate- to high-interval intensity cycling exercises), the exercises performed two sessions per week for two months and group (C) received the hemodialysis sessions only.
Who Masked: Participant
Masking Description: single (participant)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (low- to moderate-continuous intensity cycling exercises: (Active Comparator): Patients performed aerobic exercise during dialysis using Pedal machine at low- to moderate continuous intensity rating from 11 to 13 on the Borg scale for 15-30 minutes.
  warming up and cool down (approximately 10 minutes) in form of free active exercise of the lower extremities
  Interventions: Other: low- to moderate-continuous intensity cycling exercises:
- Group B (moderate- to high-interval intensity cycling exercises), (Active Comparator): Patients performed aerobic exercise during dialysis using Pedal machine at moderate-to-high interval intensity rating from 12 to 15 on the Borg scale for 15-30 minutes.
  warming up and cool down (approximately 10 minutes) in form of free active exercise of the lower extremities
  Interventions: Other: moderate- to high-interval intensity cycling exercises
- group (C) (Sham Comparator): received the hemodialysis sessions only.
  Interventions: Other: hemodialysis sessions only

INTERVENTIONS:
Other: low- to moderate-continuous intensity cycling exercises: — aerobic exercise during dialysis using Pedal machine at low- to moderate continuous intensity rating from 11 to 13 on the Borg scale for 15-30 minutes.
  warming up and cool down (approximately 10 minutes) in form of free active exercise of the lower extremities
  Other Names: low- to moderate-continuous aerobic exercise
  Arms: Group A (low- to moderate-continuous intensity cycling exercises:
Other: moderate- to high-interval intensity cycling exercises — aerobic exercise during dialysis using Pedal machine at moderate-to-high interval intensity rating from 12 to 15 on the Borg scale for 15-30 minutes.
  warming up and cool down (approximately 10 minutes) in form of free active exercise of the lower extremities
  Arms: Group B (moderate- to high-interval intensity cycling exercises),
Other: hemodialysis sessions only — hemodialysis sessions only
  Arms: group (C)

SUMMARY:
Chronic kidney disease has emerged as one of the leading causes of mortality worldwide, and it is one of a small number of non-communicable diseases that have shown an increase in associated deaths over the past 2 decades. The high number of affected individuals and the significant adverse impact of chronic kidney disease should prompt enhanced efforts for better prevention and treatment.

Chronic kidney disease is a serious medical problem, as it is associated with high risks of complications which lead to poor quality of life and physical capacity.

DETAILED DESCRIPTION:
Sixty-seven patients undergoing haemodialysis randomly be allocated into three groups, (A, B & C). Group A (low- to moderate-continuous intensity cycling exercises, group B (moderate- to high-interval intensity cycling exercises), the exercises performed two sessions per week for two months and group (C)Twenty three patients received the hemodialysis sessions only.

Group A (low- to moderate-continuous intensity cycling exercises:

Twenty three patients performed aerobic exercise during dialysis using Pedal machine at low- to moderate continuous intensity rating from 11 to 13 on the Borg scale for 15-30 minutes.

warming up and cool down (approximately 10 minutes) in form of free active exercise of the lower extremities.

Group B (moderate- to high-interval intensity cycling exercises), Twenty one patients performed aerobic exercise during dialysis using Pedal machine at moderate-to-high interval intensity rating from 12 to 15 on the Borg scale for 15-30 minutes.

warming up and cool down (approximately 10 minutes) in form of free active exercise of the lower extremities.

Inclusion Criteria:

1. Sixty seven patients of both sexes
2. Age will range from 35-55 years old.
3. BMI will be from 25-34.5 Kg/m2.
4. All patients with stage 5 of CRF.
5. All patients are stable on dialysis for at least six months before the study.
6. Stable medical and clinical hemodynamic state.

Exclusion criteria:

1. Patients with hearing impairment or mental disorder.
2. Patients with unstable angina, uncontrolled cardiac arrhythmia, decompensated heart failure, persistent systolic blood pressure (BP) greater than 200 mmHg, persistent diastolic BP greater than 120 mmHg, acute pericarditis or myocarditis.
3. Patients with auto-immune diseases.
4. Chronic inflammatory orthopedic disorders and rheumatoid arthritis.
5. Patients with history of neuromuscular disease (muscular dystrophy, myasthenia gravis, myopathy, multiple sclerosis and peripheral neuropathy).
6. Patients with chronic obstructive lung disease, restrictive lung disease or chronic chest infection.
7. Patients with BMI > 35Kg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty-seven patients of both sexes
2. Age will range from 35-55 years old.
3. BMI will be from 25-34.5 Kg/m2.
4. All patients with stage 5 of CRF.
5. All patients are stable on dialysis for at least six months before the study.
6. Stable medical and clinical hemodynamic state.

Exclusion Criteria:

* 1. Patients with hearing impairment or mental disorder. 2. Patients with unstable angina, uncontrolled cardiac arrhythmia, decompensated heart failure, persistent systolic blood pressure (BP) greater than 200 mmHg, persistent diastolic BP greater than 120 mmHg, acute pericarditis or myocarditis.

  3. Patients with auto-immune diseases. 4. Chronic inflammatory orthopedic disorders and rheumatoid arthritis. 5. Patients with history of neuromuscular disease (muscular dystrophy, myasthenia gravis, myopathy, multiple sclerosis and peripheral neuropathy).

  6. Patients with chronic obstructive lung disease, restrictive lung disease or chronic chest infection.

  7. Patients with BMI > 35Kg/m2.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Kidney Disease Quality of Life Questionnaire -SF36(KDQoL-SF36) | pre and post treatment after 2 months
  The KDQOL™-36 contains 5 subscales: The Physical Component Summary (PCS), Mental Component Summary (MCS), Burden of Kidney Disease (BKD), Symptoms and Problems of Kidney Disease (SPKD), and Effects of Kidney Disease (EKD). The first 2 subscales are a generic measure of HRQOL (and are identical to the SF-12), whereas the last 3 assess issues specific to patients with ESRD or earlier stages of chronic kidney disease.

SECONDARY OUTCOMES:
blood urea, serum creatinine | pre and post treatment after 2 months
  Blood samples are drawn from the arterial side of the hemodialysis access immediately prior to hemodialysis. Blood sample must be drawn before dialysis is started to prevent this sample from reflecting any impact of dialysis. pre and post kitz blood samples were sent to benha university hospital laboratory for estimating blood urea and creatinine.
6-min walk distance | pre and post treatment after 2 months
  6min walk test carried out before and after the intervention to determine patient physical functional capacity. According to the American Thoracic Society ,Guidelines for the Six-Minute Walk Test (ATS .2002).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy - Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Pei G, Tang Y, Tan L, Tan J, Ge L, Qin W. Aerobic exercise in adults with chronic kidney disease (CKD): a meta-analysis. Int Urol Nephrol. 2019 Oct;51(10):1787-1795. doi: 10.1007/s11255-019-02234-x. Epub 2019 Jul 22. PMID 31332699
- [Background] Wulczyn KE, Zhao SH, Rhee EP, Kalim S, Shafi T. Trajectories of Uremic Symptom Severity and Kidney Function in Patients with Chronic Kidney Disease. Clin J Am Soc Nephrol. 2022 Apr;17(4):496-506. doi: 10.2215/CJN.13010921. Epub 2022 Mar 4. PMID 35246460